CLINICAL TRIAL: NCT05157308
Title: A Cross Sectional Study for Determining Prevalence of Sarcopenia and Myosteatosis in Cirrhotic Patients and to Study the Association Between Imaging and Clinical Parameters
Acronym: Myo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Clinical Professor, Asian Institute of Gastroenterology, India
Other Study IDs: CIRR
Record Dates: First submitted 2021-11-29; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cirrhosis is associated with a wide variety of metabolic changes in the body. Ascites, hepatic encephalopathy, variceal bleeding, renal dysfunction, and hepatocellular carcinoma are the most widely recognised complications in cirrhosis. Malnutrition and muscle wasting (sarcopenia) constitute common complications, which are generally overlooked, but which negatively impact the survival, quality of life, and response to stressors like infections, sepsis and surgery in cirrhotic patients.

Cirrhotic patients with sarcopenia and myosteatosis have a higher risk of overt hepatic encephalopathy and hyperammonemia.1 It has also been shown that the patients with sarcopenia have a lower overall survival than those without sarcopenia.

The aim of the current study is to study the prevalence of myosteatosis and sarcopenia in cirrhotic patients, and to compare the clinical and anthropometric parameters for sarcopenia and myosteatosis to that of imaging parameters (CT based diagnosis).

We hypothesize that myosteatosis and sarcopenia can be estimated better with the use of CT scan as compared with clinical assessment and hence, may help in early diagnosis of these conditions.

DETAILED DESCRIPTION:
All the patients of liver cirrhosis who attend the Liver clinic of the hospital will undergo a thorough history and examination. After strict inclusion-exclusion criteria patients will be included in the study. All routine investigations required to establish the etiology of cirrhosis and to evaluate the stage of cirrhosis (Child-Turcotte-Pugh status and MELD score) would be done.

The patient will be assessed for the following anthropometric measurements -

1. Body mass index (BMI) will be calculated. In patients with Ascites- Dry body weight (kg) will be taken by- Post-paracentesis weight (kg) recorded before fluid retention (if available). OR Subtracting a percentage of weight based upon the severity of ascites (Mild Ascites- 5%, Moderate- 10%, Severe- 15%) with an additional 5% subtracted if bilateral pedal oedema is present.
2. Mid- arm circumference (MUAC) - is the circumference of the left upper arm, measured at the mid-point between the tip of the shoulder and the tip of the elbow (olecranon process and the acromium). Normal value is 29.3 in males and 28.5 mm in females.
3. Triceps Skin fold thickness - assessed in the mid arm using skin fold callipers. Normal values in adults are usually 12.5 mm in males and 16.5 mm in female.
4. Mid-arm Muscle circumference (MAMC) - defined as (mid arm circumference - triceps skin fold) x 0.314. Normal values in are 25.3 mm and 23.2 mm in adult males and females respectively.

The patients will be assessed for the indicators of muscle strength by-

1. 6 min walk Test - It measures the distance that patients can quickly walk in a flat, hard surface within 6 minute. Values > 300 m in 6 min is considered normal, while < or equal to 300 is considered low endurance while < 250m indicates frailty.
2. Balancing test - It is measured as the number of seconds that the subject can balance in three positions (feet placed side-to-side, semi-tandem, and tandem) for a maximum of 10 seconds each. The duration is recorded for each.
3. Five times sit to stand test - The subject is to sit in the chair with arms crossed over his/her chest and then to stand up as quickly as possible safely, five times without using his/her arms. Normal person should be able to do it within 12 seconds.
4. Hand Grip test - It is a function of skeletal muscle contractile strength. It would be tested using a hand held dynamometer and the average of three readings the subject's dominant hand would be taken. The same would be compared with the normative data for the age and sex of the patient.
5. Short physical performance battery - which consists of timed repeated chair stands, balance testing, and a timed 13-ft walk
6. Liver frailty index - calculated based upon HG, and balancing test.

After the anthropometric and bedside maneuvers, patient will be subjected to plain Computed tomographic (CT) scan of abdomen. CT image analysis at the L3 vertebra is almost universally recognised as a specific method to quantify muscle loss. It will be done to assess the degree of sarcopenia and myosteatosis as per the criteria.

* Total cross sectional area cm2 of abdominal skeletal muscle normalized to height = skeletal muscle index ( cm2/m2)
* Cut off for sarcopenia: 50 cm2/m2 (male) and 39 cm2/m2 (Female) It has been established to have an independent association with pooled transplantation mortality - HR : 1.84 independent of MELD.
* Cut-off for myosteatosis will be taken as Skeletal muscle radiation attenuation (SM-RA) <41 HU for patients with a body mass index [BMI] up to 24.9 kg/m2 and <33 HU for patients with a BMI ≥25 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of cirrhosis Between 18 yrs to 70 yrs attending the liver clinic of the Institute
* Those giving written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Patients with known neurological disorders or musculoskeletal disorders which can hamper the performance of physical tests
* Patients with history of neoplasia
* Patients who are unable to understand study protocol or not willing for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size required is 385 patients with 80% power and 0.05 type 1 error.
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
To compare the clinical assessment for sarcopenia (by anthropometric methods and muscle strength indicators) to that of imaging based assessment (CT based assessment) | 12 months
  The patient will be assessed for the following anthropometric measurements -2. Mid- arm circumference, Triceps Skin fold thickness (width in cms), Mid-arm Muscle circumference

SECONDARY OUTCOMES:
To determine the prevalence of sarcopenia and myosteatosis in patients with cirrhosis | 12 months
  The patients will be assessed for the indicators of muscle strength by 6 min walk Test (distance in metres), 2. Balancing test (height in cms) ,Five times sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Mithun Dr Sharma, MBBS MD DM, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana, India